CLINICAL TRIAL: NCT00068029
Title: A Randomized, Parallel Group, Three-Arm Study To Evaluate Treatment With A Combination Of Pegvisomant Plus Sandostatin Lar, Pegvisomant (Alone), And Sandostatin Lar (Alone) In Patients With Acromegaly
Brief Title: Pegvisomant And Sandostatin LAR Combination Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEGA-0435-005; A6291006
Record Dates: First submitted 2003-09-04; First posted 2003-09-05 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

INTERVENTIONS:
Drug: Pegvisomant/ Sandostatin LAR
Drug: Sandostatin LAR
Drug: Pegvisomant

SUMMARY:
The purpose of this study is to compare the safety and tolerability of combination therapy with Sandostatin LAR plus Pegvisomant to that of Sandostatin LAR alone or Pegvisomant alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acromegaly
* Received previous radiation and/or surgical treatment for their GH (Growth Hormone) producing pituitary adenoma and have required medical therapy due to failure to normalize GH (Growth Hormone) and/or IGF-I as a result of their primary treatment
* Patients that been receiving Sandostatin LAR for a minimum of 6 months prior to enrollment

Exclusion Criteria:

* Presence of other conditions that may result in abnormal GH (Growth Hormone) and/or IGF-I concentrations
* Patients on current medical therapy other than Sandostatin LAR
* AST/ALT >= 3xULN (upper limits of normal)
* Pituitary adenoma within 3mm of optic chiasm confirmed by recent MRI
* Visual field defects (except post-surgical stable residual defects)
* Unable to self administer drug
* Radiotherapy within 12 months of entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2003-10; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing treatment-emergent adverse events across the duration fo the study

SECONDARY OUTCOMES:
Percentage of patients with normalization of IGF-I, at Week 40, in the two randomized groups (Sandostatin LAR plus pegvisomant and pegvisomant alone). Normal IGF-I is defined as a value within the normal reference range for age for the study specific

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- United States (4):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Charlottesville, Virginia
- Australia (3):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Fitzroy, Victoria
  - Pfizer Investigational Site, Fizroy, Victoria
- Brazil (2):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, SÃ£o Paulo, São Paulo
- Canada (2):
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Toronto, Ontario
- France (2):
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nice
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Hanover
- Italy (4):
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Torino
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Col La Raza, Mexico DF
- Pfizer Investigational Site, Nijmegen, Netherlands
- Pfizer Investigational Site, Oslo, Norway
- Spain (2):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
- United Kingdom (5):
  - Pfizer Investigational Site, Belfast, Antrim
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Oxford

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=PEGA-0435-005&StudyName=Pegvisomant+And+Sandostatin+LAR+Combination+Study